Study of the Efficacy of GGON: a Cognitive Training App for Orthorexia Nervosa Module.

NCT06288347 18/04/2022

## **INFORMED CONSENT**

Informed Consent (38325) Description: The research project for which we are asking your participation is entitled: "Validation of the GGON App". In order for you to participate in this study, it is necessary to have your consent, and that you know the basic information so that such consent can be considered truly informed. Therefore, please read the following information carefully. Before accepting the text, if you have any doubts, you can contact the principal investigator of the project, by telephone or by e-mail below. The basic information you should know is as follows: a) Aim of the study: To analyze the effectiveness of the GGON App. b) Methodology to be used for the study, type of collaboration expected from you and duration of such collaboration: You will be asked to complete a series of questionnaires that will take approximately 10 minutes to complete. c) Possible discomforts and risks of your participation in the study: Participation does not involve any risk. However, some people may feel uncomfortable answering certain questions about their diet and behavior. d) Measures to ensure adequate compensation in case you suffer any harm: The person will be offered face-to-face or videoconference contact in order to deal with the harm caused, and if necessary, referral to a professional. e) Expected benefits of the research: It is expected to learn about the effectiveness of the App in order to expand its use. f) Consequences of non-participation: The decision not to participate will not affect your right to health care, nor the relationship with the people who proposed you to participate, which will be just as cordial and dedicated with those who refuse to participate as with those who do participate. g) Possibility of withdrawal at any time and consequences: If you respond to the questions proposed to you, it is tacitly understood that you have understood the objective of this study, that you have been able to ask and clarify any doubts that may have been initially raised and that you agree to participate in the study. However, only surveys that have been fully completed will be taken into account. Thus, the partial results of the surveys will be discarded. h) Who has financed the study: The Generalitat Valenciana through the grant for emerging research groups (GVA/2021/162). i) Which institution is carrying out the study: The Universitat de València. j) Free of charge for participation: Participants will not obtain any financial compensation for their participation in this study. k) Expected subsequent use of the results: The results will be used for teaching, research and/or scientific publication purposes. 1) Research Team: Principal Investigator: María Roncero Sanchis, Martha Giraldo, Juan Ramón Barrada and Guy Doron. With the collaboration of Marta Corberán Vallet. m) Principal investigator's contact information for clarifications or queries: María Roncero Sanchis. Av. Blasco Ibáñez, 21. Faculty of Psychology. Dept. of Personality, Evaluation and Psychological Treatments. POSTAL CODE: 46010. Valencia. Valencia, Spain. Email: maria.roncero@uv.es. Telf: 963983364. n) The project will be carried out following the international ethical criteria contained in the Declaration of Helsinki. 2.- CONFIDENTIALITY COMMITMENT. a) Measures to ensure respect for privacy and confidentiality of personal data: Appropriate measures

have been taken to ensure complete confidentiality of personal data of experimental subjects participating in this study, in accordance with the Law of Protection of Personal Data (LOPD) 3/2018, of December 5. b) Measures to access information relevant to you arising from the research or from the overall results: You have the right to access the information generated in the study, although because it is anonymous data you will not be given specific information about your results. You can send an-e-mail to the principal investigator to request the general results. c) Measures taken because it is an anonymized study: An effective anonymization system has been established that does not allow subsequent identification of the individual. In the use made of the results of the study, for teaching, research and/or publication purposes, due anonymization of personal data will always be respected, so that the research subjects will not be identified or identifiable.